CLINICAL TRIAL: NCT06210776
Title: A Multi-center Prospective Observational Study to Assess the Effectiveness and Safety of Trastuzumab Deruxtecan in Chinese Breast Cancer Patients (REFRESH)
Brief Title: A Study to Assess the Effectiveness of Trastuzumab Deruxtecan in Chinese Breast Cancer Patients (REFRESH)
Status: Recruiting | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: DSCN-EHT-NIS-BC002
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: HER2-positive Breast Cancer; HER2-low Breast Cancer; Breast Cancer; Advanced Cancer
Keywords: HER2-positive breast cancer; HER2-low breast cancer; Breast cancer; Advanced cancer; Unresectable or metastatic breast cancer; Trastuzumab deruxtecan; T-DXd
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Patients with unresectable or metastatic HER2+ breast cancer who have received one or more prior anti-HER2-based regimens.
  Interventions: Drug: Trastuzumab deruxtecan
- Cohort B: Patients with unresectable or metastatic HER2-low breast cancer patients who have received at least a prior systemic therapy in the metastatic setting or developed disease recurrence during or within 6 months of completing adjuvant chemotherapy.
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Intravenous infusion
  Other Names: T-DXd

SUMMARY:
This multi-center observational prospective study will collect real-world clinical and patient-reported outcome data from eligible patients with unresectable or metastatic HER2+ breast cancer who have received one or more prior anti-HER2-based regimens or patients with unresectable or metastatic HER2-low (IHC 1+ or IHC 2+, ISH-) breast cancer who have received at least a prior systemic therapy in the metastatic setting, or developed disease recurrence during or within 6 months of completing adjuvant chemotherapy.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate real-world time to next treatment or date of death from index date (T-DXd treatment initiation date)(rwTTNT) in each cohort. The secondary objectives of this study are to describe treatment patterns in eligible patients with HER2+ or HER2-low unresectable or mBC who are newly initiating T-DXd in a real-world setting, to describe demographic and clinical characteristics, to assess the safety and tolerability through the collection of physician-reported SEIs, to characterize the management of SEIs, to evaluate real-world time to treatment discontinuation (rwTTD) of T-DXd, and to evaluate patient-reported tolerability.

This decision to treat the patient with T-DXd will be made prior to, and independent of, their participation in this study. Eligible patients willing to participate will be enrolled consecutively in the study and followed up from index date (T-DXd treatment initiation date) until end of study, death, or withdrawal of consent, or loss to follow-up (LTFU), or study closure, whichever occurs first.

ELIGIBILITY:
Patients must meet all of the following inclusion criteria to be eligible for the study:

1. ≥18 years of age at time of consent.
2. Pathologically documented breast cancer that is unresectable or metastatic.
3. Cohort A: Patients with confirmed HER2+ (IHC 3+ or IHC2+, ISH+); and patients have received one or more prior anti-HER2-based regimens; and patients should have received no more than 2 lines therapy in the metastatic settings.

   Cohort B: Patients with confirmed HER2-low expression (IHC 1+ or IHC 2+, ISH-); and patients have received at least a prior systemic therapy in the metastatic setting or developed disease recurrence during or within 6 months of completing adjuvant chemotherapy; and patients should have received no more than 2 lines of previous chemotherapy regimen in the metastatic settings.
4. Decision to newly initiate T-DXd or just have started the first dose no longer than 14 days after the index date per approved label in China.
5. Capable of providing informed consent.
6. Patients capable of completing questionnaires are preferred. If the participant is unable to complete the questionnaire (e.g., being blind, illiterate, not fluent in the available language, or ePRO system is not ready), that participant is exempted from completing PRO questionnaires but may still participate in the study.

Patients who meet any of the following criteria will be excluded from the study:

1. Pregnancy or breastfeeding.
2. Patients who at time of data collection for this study are participating in or have participated in an interventional study that remains blinded.
3. Patients who have known to have hypersensitivity reactions to the active substance of T-DXd or any excipients.
4. Patients who have been judged by the investigator to be unfit to participate the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 800 eligible subjects with HER2+ or HER2-low unresectable or mBC will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Real World Time to Next Treatment (rwTTNT) in Participants With HER2-positive and HER2-low Unresectable or Metastatic Breast Cancer | Assessed over a 36-month period
  Time to next treatment or death from index date will be assessed.

SECONDARY OUTCOMES:
Change in T-DXd Dosing in Participants With HER2-positive and HER2-low Unresectable or Metastatic Breast Cancer | Assessed over a 36-month period
Duration of Treatment (DoT) in Participants With HER2-positive and HER2-low Unresectable or Metastatic Breast Cancer | Assessed over a 36-month period
  Duration of treatment is defined as the length of time a patient is treated.
Change in Dose Amendment in Participants With HER2-positive and HER2-low Unresectable or Metastatic Breast Cancer | Assessed over a 36-month period
Percentage of Participants With HER2-positive and HER2-low Unresectable or Metastatic Breast Cancer, Based on Demographic and Clinical Characteristics | Assessed over a 36-month period
Number of Participants Reporting Physician-reported Safety Events of Interest (SEI) in Participants With HER2-positive and HER2-low Unresectable or Metastatic Breast Cancer | Assessed over a 36-month period
Number of Participants Reporting Prophylactic and Reactive Treatment for SEI Management | Assessed over a 36-month period
Real-world Time to Discontinuation (rwTTD) in Participants With HER2-positive and HER2-low Unresectable or Metastatic Breast Cancer | Assessed over a 36-month period
  Time to discontinuation is defined as time from index date to the earliest date of T-DXd discontinuation, or date of death.
Change in Patient's Global Impression of Treatment Tolerability in Participants With HER2-positive and HER2-low Unresectable or Metastatic Breast Cancer | Baseline up to 1 month post-T-DXd treatment
Number of Participants Reporting Symptom Items From National Cancer Institute Patient Reported Outcome Common Terminology Criteria for Adverse Events | Baseline up to 1 month post-T-DXd treatment
Number of Participants Reporting Nausea and Vomiting Based on Symptom Diary Data | Baseline up to 1 month post-T-DXd treatment

CONTACTS AND LOCATIONS:
Overall Officials: Director, Study Director — Daiichi Sankyo China
Locations (54):
- China (54):
  - China-Japan Friendship Hospital, Beijing
  - Peking University First Hospital, Beijing
  - The Fifth Medical Center of the Chinese PLA General Hospital, Beijing
  - Peking University Shougang Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing GoBroad Hospital, Beijing
  - Sichuan Cancer Hospital, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - Affiliated Zhongshan Hospital of Dalian University, Dalian
  - The First People's Hospital of Foshan, Foshan
  - Fujian Cancer Hospital, Fuzhou
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - Hainan Cancer Hospital, Haikou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Provincial Cancer Hospital, Hefei
  - Jiamusi Cancer Hospital, Jiamusi
  - Yunnan Cancer Hospital, Kunming
  - The First People's Hospital of Lianyungang, Lianyungang
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang
  - Jiangxi Cancer Hospital, Nanchang
  - Nanchang Third Hospital, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - The Peoples of Guangxi Zhuang Autonomous Region, Nanning
  - Affiliated Hospital Of Nantong University, Nantong
  - Ningbo No.2 Hospital, Ningbo
  - Qingdao Central Hospital, Qingdao
  - Fudan University Shanghai Cancer Center, Shanghai
  - Changhai Hospital, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - Liaoning Cancer Hospital & Institute, Shenyang
  - The University of Hong Kong- Shenzhen Hospital, Shenzhen
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen
  - Shanxi Provincial Cancer Hospital, Taiyuan
  - Tangshan People's Hospital, Tangshan
  - Tianjin Cancer Hospital Airport Hospital, Tianjin
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi
  - Weifang People's Hospital, Weifang
  - Wenzhou Central Hospital, Wenzhou
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Xi'an International Medical Center Hospital, Xi'an
  - The First Affilital of Xiamen University, Xiamen
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - General Hospital of Ningxia Medical University, Yinchuan
  - Henan Cancer Hospital, Zengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Henan Provincial People's Hospital, Zhengzhou
  - Zhongshan City People's Hospital, Zhongshan
  - The Fifth Affiliated Hospital, Sun Yat-sen University, Zhuhai

IPD SHARING:
Plan to Share IPD: No